CLINICAL TRIAL: NCT00358774
Title: A Double-blind, Placebo-controlled Trial to Test the Efficacy of Homeopathic Nasal Formulation for the Management of Experimental Rhinoviral Colds in an Outpatient Setting
Brief Title: Efficacy of Homeopathic Nasal Formulation for Management of Experimental Rhinoviral Colds
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2001-089
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Common Cold
Keywords: homeopathic; common cold; Research Subjects
MeSH Terms: conditions — Common Cold

INTERVENTIONS:
Procedure: homeopathic nasal spray

SUMMARY:
Common colds affect many people and are the cause of bothersome symptoms such as runny or stuffy nose, sore throat, headache and sneezing. Common colds can also cause more severe illnesses in certain groups of people like the elderly, people with chronic lung diseases such as asthma.

This study is designed to test whether a non-drug (homeopathic) nasal spray will reduce the incidence of colds, decrease cold related symptoms or shorten the length of the cold.

DETAILED DESCRIPTION:
Common colds are the most frequent type of respiratory infection, and although the clinical manifestations are usually not life threatening or debilitating, they cause annoying symptoms such as nasal congestion, rhinorrhea, malaise, sore throat and sneezing, that can interfere with activities of daily living. Furthermore, colds can cause more severe illnesses in certain people including: infants, the elderly, and people with asthma, chronic lung diseases, or immune deficiency.

This clinical trial is designed to test whether a new homeopathic formulation has beneficial effects on the management of common colds that have been induced by inoculation of rhinovirus into the nose of healthy subjects.

The objective of this research clinical study is to evaluate the effectiveness of a homeopathic nasal formulation for the management of experimentally-induced common colds as indicated by a reduction in:

* Cold incidence compared to placebo,
* Symptom severity compared to placebo
* Cold duration compared to placebo
* Infection rate compared to placebo
* Duration of virus shedding compared to placebo or
* Amount of virus shedding compared to placebo

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible for enrollment into this study, subject must:

1. Be healthy based on medical history, physical and nasal examination
2. Be male or non-pregnant, non-lactating female (women of child-bearing potential must be using an acceptable form of contraception, including abstinence, as determined by the Investigator)
3. Be between 18 - 60 years old
4. Be willing to refrain from taking nasal decongestants, antihistamines or cough/cold preparations (this includes dietary supplements and homeopathic preparations used specifically for cold/flu e.g., vitamin C, zinc, echinacea) within the 7 days prior to Day 0 and through Day 5
5. Be willing to refrain from taking any other medication (except contraceptive preparations, hormone replacement therapy, acne medication) within 2 days prior to Day 0 and through Day 5
6. Has read, signed and received a copy of the Informed Consent Form.

Exclusion Criteria:

Subjects will be excluded from the study if they:

1. Are intolerant of nasal sprays
2. Require a medication on regular basis (3 or more times/week) except contraceptive preparations, hormone replacement therapy, acne medication
3. Have a history of chronic diseases such as respiratory (e.g., chronic rhinitis, sinusitis, asthma, chronic bronchitis, pneumonia, persistent or chronic cough, emphysema, breathing problems, excessive phlegm or mucus), cardiovascular, endocrine, neurological, hepatic, gastrointestinal, renal, hematological, urological, immunological, ophthalmic diseases requiring medication
4. Have a history of headache (e.g., frequent migraines, cluster headaches, 3+ headaches/week)
5. Have had cold symptoms in the past 14 days
6. Are currently symptomatic with respiratory allergy
7. Have any clinically significant abnormalities of the upper (including history of nose bleeds, nasal abnormalities or other nasal pathology such as irreversible nasal mucosal hypertrophy or severe nasal septal deviation) or lower respiratory tract
8. Have used any investigational medication in the past 30 days
9. Are smokers
10. Have serum neutralizing antibody titer of >1 to RV16 at Pre-screening
11. Have a condition or is taking a medication that the Investigator and/or designee believes could jeopardize the safety of the subject, would interfere with the evaluation or confound the interpretation of the study results
12. Have positive urine pregnancy test (for female subjects only)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Start 2001-03; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects who become infected and show the presence of a cold.(active vs placebo)

SECONDARY OUTCOMES:
The proportion of subjects who become infected.
The mean number of days that virus was shed for inoculated subjects (active vs placebo)

CONTACTS AND LOCATIONS:
Overall Officials: James E Gern, MD, Principal Investigator — University of Wisconsin, Madison